CLINICAL TRIAL: NCT05253638
Title: Evaluation Of Serum MIF Level in SLE Patients and It's Association With Disease Activity and Severity
Brief Title: Evaluation Of Serum MIF Level in SLE Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Manal Kamal, Principal investigator, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MIF S
Record Dates: First submitted 2021-11-28; First posted 2022-02-24 (Actual); Last update posted 2022-02-24 (Actual); Status verified 2022-02

CONDITIONS: Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- study group (Experimental): Patients will be recruited from the Rheumatology, Rehabilitation Department from The in patient and out patient clinic of Assiut University Hospitals with an informed consent will be obtained from all patients.
  Adult SLE patients >18 who fulfilled the 2012 systemic lupus international collaborating clinics (SLICC) criteria
  Interventions: Diagnostic Test: Macrophage migration inhibitory factor

INTERVENTIONS:
Diagnostic Test: Macrophage migration inhibitory factor — Assessment of disease activity: This assessment will be performed using the systemic lupus erythematosus disease activity index (SLEDAI). The SLEDAI is an index designed to assess disease activity in the preceding 10 days, with 24 weighted clinical and laboratory variables corresponding to 9 different organs/systems. The SLEDAI score ranges from 0 to 105 Renal activity will be evaluated with the renal-SLEDAI (rSLEDAI), which represents the sum of the renal items of the SLEDAI. The rSLEDAI includes the following items: proteinuria, pyuria, erythrocyturia, and urine casts; each one is scored with 0 meaning absence or 4 points meaning presence; therefore, the maximum rSLEDAI is 16
  Other Names: Macrophage migration inhibitory factor (MIF)

SUMMARY:
Systemic lupus erythematosis (SLE) is a chronic autoimmune disease characterized by production of autoantibodies and the deposition of immune complexes, affecting a wide range of organs. The clinical onset of SLE derives from the interaction between genetic predisposition and environmental, immunological and hormonal factors, with a strong predilection for women of childbearing age.

SLE is usually diagnosed in young women in the third decade of life and represents the leading cause of systemic disease with secondary kidney involvement. Lupus nephritis (LN) occurs in ~50% of patients with SLE and is the most common, but not the only, cause of kidney injury in SLE. LN typically develops early in the disease course, generally within the first 6 to 36 months, and may be present at initial diagnosis.

Macrophage migration inhibitory factor (MIF) is a pleiotropic inflammatory cytokine with regulatory roles in innate and adaptive immunity and is implicated in the pathogenesis of autoimmune diseases including SLE.

MIF actively participates in multiple stages of the inflammatory response, acting on cells directly and/or potentiating the effects exerted by other stimuli. MIF overcomes the inhibitory effects of glucocorticoids on TNF alpha, IL-1 beta, IL-6, and IL-8 production.

MIF is implicated in the pathogenesis of other autoimmune diseases including rheumatoid arthritis (RA), type 1 diabetes, multiple sclerosis and Guillain Barré syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Adult SLE patients >18 years
* fulfilled the 2012 systemic lupus international collaborating clinics (SLICC) criteria

Exclusion Criteria:

* Patients with overlap syndrome, pregnancy, active infection, diseases other than SLE that might produce abnormal proteinuria.
* Individuals with other autoimmune diseases (rheumatoid arthritis, dermatomyositis, scleroderma, mixed connective tissue disease).

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-02-22 (Estimated); Primary Completion 2022-12-22 (Estimated); Study Completion 2022-12-28 (Estimated)

PRIMARY OUTCOMES:
level of Serum Macrophage Migration Inhibitory Factor Level in Systemic Lupus Erythematosus Patients and Its Association with Disease Activity and Severity | 1 hour
  measurement through ELISA

IPD SHARING:
Plan to Share IPD: Undecided